CLINICAL TRIAL: NCT00079989
Title: A Phase 3, Open-label, Noncomparative Study of Tigecycline for the Treatment of Subjects With Selected Serious Infections Due to Resistant Gram-negative Organisms Such as Enterobacter Species, Acinetobacter Baumannii, and Klebsiella Pneumoniae
Brief Title: Study Evaluating Tigecycline in Selected Serious Infections Due to Resistant Gram-Negative Organisms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-309
Record Dates: First submitted 2004-03-19; First posted 2004-03-23 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Gram-Negative Bacterial Infections
Keywords: Bacterial Infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Bacterial Infections | interventions — Tigecycline

INTERVENTIONS:
Drug: tigecycline

SUMMARY:
To evaluate the safety and efficacy of tigecycline in the treatment of subjects with selected serious infections caused by resistant gram-negative bacteria, eg, Acinetobacter baumannii, Enterobacter species, Klebsiella pneumoniae or other resistant gram-negative pathogens, for whom antibiotics have failed or who cannot tolerate other appropriate antimicrobial therapies. The primary efficacy endpoint will be the clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older
* Isolation of a resistant gram-negative pathogen, eg, Enterobacter species, Acinetobacter baumannii, Klebsiella pneumoniae, or other resistant gram-negative pathogens, alone or as 1 isolate of a polymicrobial infection
* Resistant gram-negative organisms are defined by the likely presence of ESBL or related mechanisms which limit the therapeutic alternatives for the treatment of complicated infections

Exclusion Criteria:

* Subjects with any concomitant condition or taking any concomitant medication that, in the opinion of the investigator, could preclude an evaluation of a response or make it unlikely that the contemplated course of therapy or follow-up assessment will be completed or that will substantially increase the risk associated with the subject's participation in this study
* Anticipated length of antibiotic therapy < 7 days
* Known or suspected hypersensitivity to tigecycline or other compounds related to this class of antibacterial agents (eg, tetracyclines, minocycline, doxycycline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2003-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer